CLINICAL TRIAL: NCT07132307
Title: Reducing Obstructive Sleep Apnea After Hypoglossal Nerve Stimulation Through
Brief Title: Reducing Obstructive Sleep Apnea After Hypoglossal Nerve Stimulation Through Mandibular Advancement
Acronym: ROHMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202504015
Record Dates: First submitted 2025-07-22; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Otolaryngology; Mandibular advancement device; Hypoglossal nerve stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Pilot, single-intervention study
Masking Description: no masking required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mandibular Advancement Device (MAD) (Experimental): This study is experimental. It involves a single-intervention design where participants who have failed hypoglossal nerve stimulation (HGNS) therapy for moderate to severe obstructive sleep apnea (OSA) will be treated with a mandibular advancement device (MAD).
  Interventions: Device: Mandibular advancement device (MAD)

INTERVENTIONS:
Device: Mandibular advancement device (MAD) — The intervention in this study involves fitting and using a mandibular advancement device (MAD), specifically the ProSomnus Sleep Device, to treat moderate to severe obstructive sleep apnea (OSA) in patients who are intolerant to CPAP and have failed hypoglossal nerve stimulation (HGNS) therapy.
  Other Names: ProSomnus Sleep Device.

SUMMARY:
The purpose of this study is to evaluate the effectiveness, feasibility, and safety of mandibular advancement devices (MAD) for treating severe obstructive sleep apnea (OSA) in patients who are CPAP intolerant and have failed hypoglossal nerve stimulation (HGNS).

DETAILED DESCRIPTION:
ROHMA is a pilot/single intervention study aiming to evaluate effectiveness of a mandibular advancement device (MAD) for treating moderate to severe obstructive sleep apnea (OSA) in patients who have failed hypoglossal nerve stimulation therapy (HGNS). Individuals who received a HGNS therapy at Washington University from April 4 2019 to October 20 2024, or were enrolled in a prior study (HRPO #: 202309014) will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Ability to read, write, speak, and understand English.
* Failure of hypoglossal nerve stimulation (HGNS) therapy, defined as intolerance to HGNS or insufficient AHI reduction based on modified Sher criteria while using HGNS.
* Ability to insert and remove the mandibular advancement device (MAD) independently.
* Ability to complete all study assessments and evaluations, including home sleep apnea tests (HSAT).
* Ability to abstain from any other treatment for obstructive sleep apnea (OSA) during the entire study duration.
* Access to an internet-connected device (phone, tablet, or laptop) with a camera.

Exclusion Criteria:

* Age over 70 years.
* Inability to use a mandibular advancement device (MAD), defined as having fewer than 9 healthy teeth per dental arch.
* Prior intolerance to MAD therapy.
* Previous participation in a trial involving the use of oral appliances.
* Chronic nasal obstruction.
* Dependence on or frequent use of medications that alter consciousness, respiration, or alertness.
* Insomnia and/or use of medications to treat insomnia.
* Sleep disorders such as narcolepsy, insomnia, restless leg syndrome, or other disorders affecting sleep, and/or use of medications to treat such disorders.
* Substance abuse.
* Unstable psychiatric disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders | through study completion on average 8 weeks
  The proportion of responders will be defined as number of participants with more than a 50% reduction in apnea-hypopnea index (AHI) and a final AHI less than 15 (modified Sher criteria) after treatment compared to baseline, divided by the total number of participants treated with mandibular advancement device.
  The AHI is a standardized index used to diagnose and determine the severity of sleep apnea. AHI will be obtained from a home sleep apnea test completed by the participants and reviewed by a trained sleep neurologist.

SECONDARY OUTCOMES:
Magnitude of change in apnea-hypopnea index (AHI). | through study completion on average 8 weeks
  The magnitude of change in apnea-hypopnea index (AHI) refers to the difference in AHI values measured before and after using the mandibular advancement device (MAD).
Change in Oxygen desaturation index (ODI) | through study completion on average 8 weeks
  The ODI is an index used to measure the degree of oxygen desaturation during sleep. The ODI will be obtained from the sleep study results by a trained sleep neurologist.
  Change in ODI will be calculated as the difference ODI pre and post treatment sleep studies.
Change in the time spent below oxygen saturation 90% | through study completion on average 8 weeks
  The time spent below oxygen saturation 90% difference will be defined as the difference of the length of time where participants have an arterial saturation of oxygen below 90% during pre- and post- treatment sleep study.
Changes in the mean arterial oxygen saturation (SaO2) | through study completion on average 8 weeks
  The changes in arterial oxygen saturation (SaO2) will be defined as the difference in the mean arterial oxygen saturation recorded during pre- and post- treatment sleep studies.
Adherence to MAD use | through study completion on average 8 weeks
  Adherence is defined as using the MAD for at least 4 hours per night on at least 5 out of 7 nights during the entire intervention period.
  The proportion of participants meeting this adherence criterion is calculated and reported to assess feasibility and compliance with the treatment.
Change in Epworth Sleepiness Scale (ESS) | through study completion on average 8 weeks
  The Epworth Sleepiness Scale (ESS) is measured by asking participants to rate their likelihood of falling asleep in eight different everyday situations on a scale from 1 (least likely) to 7 (most likely).
  The total ESS score reflects the level of daytime sleepiness, with higher scores indicating greater sleepiness.
  Change in the Epworth Sleepiness Scale (ESS) is assessed by comparing participants' ESS scores before starting mandibular advancement device (MAD) therapy (baseline) with their scores after the intervention period.
Epworth Sleepiness Scale (ESS) improvement | through study completion on average 8 weeks
  The Epworth Sleepiness Scale (ESS) is measured by asking participants to rate their likelihood of falling asleep in eight different everyday situations on a scale from 1 (least likely) to 7 (most likely).
  The total ESS score reflects the level of daytime sleepiness, with higher scores indicating greater sleepiness.
  Change in the Epworth Sleepiness Scale (ESS) is assessed by comparing participants' ESS scores before starting mandibular advancement device (MAD) therapy (baseline) with their scores after the intervention period.
  The proportion of participants with improved ESS will be calculated as number of participants whose ESS score changes exceed the minimal clinically important difference (MCID) of 2.4 points divided by the total number of participants.
Symptoms of Nocturnal Obstruction and Related Events (SNORE-25) | through study completion on average 8 weeks
  The Symptoms of Nocturnal Obstruction and Related Events (SNORE-25) is a validated 25-item questionnaire used to assess sleep-disorder related morbidity by capturing the frequency and severity of symptoms associated with obstructive sleep apnea. The total score ranges from 0 to 5, with higher scores indicating a greater health burden related to sleep-disordered breathing.
  Change in the Symptoms of Nocturnal Obstruction and Related Events (SNORE-25) scale is assessed by comparing participants' SNORE-25 scores before starting mandibular advancement device (MAD) therapy with their scores after completing the intervention period.
Clinical Global Impression of Improvement (CGI-I) Scale | through study completion on average 8 weeks
  The Clinical Global Impression of Improvement (CGI-I) scale is a validated, widely used tool that asks participants to rate their overall response to a treatment-in this case, mandibular advancement device (MAD) therapy for obstructive sleep apnea.
  Participants select one of seven response options: Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, or Very Much Worse. The proportion of participants reporting improvement is defined as those who choose "Much Improved" or "Very Much Improved" divided by the total number of participants completing the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skirko JR, James KT, Garrison LP, Weaver EM. Development of a Sleep Apnea-Specific Health State Utility Algorithm. JAMA Otolaryngol Head Neck Surg. 2020 Mar 1;146(3):270-277. doi: 10.1001/jamaoto.2019.4469. PMID 31999308
- [Background] Wojda M, Kostrzewa-Janicka J, Sliwinski P, Bielen P, Jurkowski P, Wojda R, Mierzwinska-Nastalska E. Mandibular Advancement Devices in Obstructive Sleep Apnea Patients Intolerant to Continuous Positive Airway Pressure Treatment. Adv Exp Med Biol. 2019;1150:35-42. doi: 10.1007/5584_2018_275. PMID 30255301
- [Background] Abbasi A, Gupta SS, Sabharwal N, Meghrajani V, Sharma S, Kamholz S, Kupfer Y. A comprehensive review of obstructive sleep apnea. Sleep Sci. 2021 Apr-Jun;14(2):142-154. doi: 10.5935/1984-0063.20200056. PMID 34381578
- [Background] Franklin KA, Lindberg E. Obstructive sleep apnea is a common disorder in the population-a review on the epidemiology of sleep apnea. J Thorac Dis. 2015 Aug;7(8):1311-22. doi: 10.3978/j.issn.2072-1439.2015.06.11. PMID 26380759
- [Background] Woo HJ, Lim JH, Ahn JC, Lee YJ, Kim DY, Kim HJ, Rhee CS, Won TB. Characteristics of Obstructive Sleep Apnea Patients With a Low Body Mass Index: Emphasis on the Obstruction Site Determined by Drug-Induced Sleep Endoscopy. Clin Exp Otorhinolaryngol. 2020 Nov;13(4):415-421. doi: 10.21053/ceo.2019.00794. Epub 2020 Apr 29. PMID 32344992
- [Background] Wong SJ, Luitje ME, Karelsky S. Patterns of Obstruction on DISE in Adults With Obstructive Sleep Apnea Change With BMI. Laryngoscope. 2021 Jan;131(1):224-229. doi: 10.1002/lary.28777. Epub 2020 Jun 8. PMID 32511760
- [Background] Lv R, Liu X, Zhang Y, Dong N, Wang X, He Y, Yue H, Yin Q. Pathophysiological mechanisms and therapeutic approaches in obstructive sleep apnea syndrome. Signal Transduct Target Ther. 2023 May 25;8(1):218. doi: 10.1038/s41392-023-01496-3. PMID 37230968
- [Background] Kazemeini E, Van de Perck E, Dieltjens M, Willemen M, Verbraecken J, Op de Beeck S, Vanderveken OM. Critical to Know Pcrit: A Review on Pharyngeal Critical Closing Pressure in Obstructive Sleep Apnea. Front Neurol. 2022 Feb 22;13:775709. doi: 10.3389/fneur.2022.775709. eCollection 2022. PMID 35273554
- [Background] Rotenberg BW, Murariu D, Pang KP. Trends in CPAP adherence over twenty years of data collection: a flattened curve. J Otolaryngol Head Neck Surg. 2016 Aug 19;45(1):43. doi: 10.1186/s40463-016-0156-0. PMID 27542595
- [Background] Aurora RN, Casey KR, Kristo D, Auerbach S, Bista SR, Chowdhuri S, Karippot A, Lamm C, Ramar K, Zak R, Morgenthaler TI; American Academy of Sleep Medicine. Practice parameters for the surgical modifications of the upper airway for obstructive sleep apnea in adults. Sleep. 2010 Oct;33(10):1408-13. doi: 10.1093/sleep/33.10.1408. PMID 21061864
- [Background] Thaler E, Schwab R, Maurer J, Soose R, Larsen C, Stevens S, Stevens D, Boon M, Huntley C, Doghramji K, Waters T, Kominsky A, Steffen A, Kezirian E, Hofauer B, Sommer U, Withrow K, Strohl K, Heiser C. Results of the ADHERE upper airway stimulation registry and predictors of therapy efficacy. Laryngoscope. 2020 May;130(5):1333-1338. doi: 10.1002/lary.28286. Epub 2019 Sep 14. PMID 31520484
- [Background] Mashaqi S, Patel SI, Combs D, Estep L, Helmick S, Machamer J, Parthasarathy S. The Hypoglossal Nerve Stimulation as a Novel Therapy for Treating Obstructive Sleep Apnea-A Literature Review. Int J Environ Res Public Health. 2021 Feb 9;18(4):1642. doi: 10.3390/ijerph18041642. PMID 33572156
- [Background] Kezirian EJ, Goding GS Jr, Malhotra A, O'Donoghue FJ, Zammit G, Wheatley JR, Catcheside PG, Smith PL, Schwartz AR, Walsh JH, Maddison KJ, Claman DM, Huntley T, Park SY, Campbell MC, Palme CE, Iber C, Eastwood PR, Hillman DR, Barnes M. Hypoglossal nerve stimulation improves obstructive sleep apnea: 12-month outcomes. J Sleep Res. 2014 Feb;23(1):77-83. doi: 10.1111/jsr.12079. Epub 2013 Sep 4. PMID 24033656
- [Background] Vanderveken OM, Maurer JT, Hohenhorst W, Hamans E, Lin HS, Vroegop AV, Anders C, de Vries N, Van de Heyning PH. Evaluation of drug-induced sleep endoscopy as a patient selection tool for implanted upper airway stimulation for obstructive sleep apnea. J Clin Sleep Med. 2013 May 15;9(5):433-8. doi: 10.5664/jcsm.2658. PMID 23674933
- [Background] Manetta IP, Ettlin D, Sanz PM, Rocha I, Meira E Cruz M. Mandibular advancement devices in obstructive sleep apnea: an updated review. Sleep Sci. 2022 Apr-Jun;15(Spec 2):398-405. doi: 10.5935/1984-0063.20210032. PMID 35371398
- [Background] Chung JW, Enciso R, Levendowski DJ, Morgan TD, Westbrook PR, Clark GT. Treatment outcomes of mandibular advancement devices in positional and nonpositional OSA patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 May;109(5):724-31. doi: 10.1016/j.tripleo.2009.11.031. Epub 2010 Mar 17. PMID 20299246
- [Background] Dieltjens M, Braem MJ, Van de Heyning PH, Wouters K, Vanderveken OM. Prevalence and clinical significance of supine-dependent obstructive sleep apnea in patients using oral appliance therapy. J Clin Sleep Med. 2014 Sep 15;10(9):959-64. doi: 10.5664/jcsm.4024. PMID 25142766
- [Background] Marklund M, Stenlund H, Franklin KA. Mandibular advancement devices in 630 men and women with obstructive sleep apnea and snoring: tolerability and predictors of treatment success. Chest. 2004 Apr;125(4):1270-8. doi: 10.1378/chest.125.4.1270. PMID 15078734
- [Background] Vecchierini MF, Attali V, Collet JM, d'Ortho MP, Goutorbe F, Kerbrat JB, Leger D, Lavergne F, Monaca C, Monteyrol PJ, Mullens E, Pigearias B, Martin F, Khemliche H, Lerousseau L, Meurice JC. Mandibular advancement device use in obstructive sleep apnea: ORCADES study 5-year follow-up data. J Clin Sleep Med. 2021 Aug 1;17(8):1695-1705. doi: 10.5664/jcsm.9308. PMID 34165074
- [Background] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Background] Rosen IM, Kirsch DB, Carden KA, Malhotra RK, Ramar K, Aurora RN, Kristo DA, Martin JL, Olson EJ, Rosen CL, Rowley JA, Shelgikar AV; American Academy of Sleep Medicine Board of Directors. Clinical Use of a Home Sleep Apnea Test: An Updated American Academy of Sleep Medicine Position Statement. J Clin Sleep Med. 2018 Dec 15;14(12):2075-2077. doi: 10.5664/jcsm.7540. PMID 30518456
- [Background] Malhotra A, Ayappa I, Ayas N, Collop N, Kirsch D, Mcardle N, Mehra R, Pack AI, Punjabi N, White DP, Gottlieb DJ. Metrics of sleep apnea severity: beyond the apnea-hypopnea index. Sleep. 2021 Jul 9;44(7):zsab030. doi: 10.1093/sleep/zsab030. PMID 33693939
- [Background] Piccirillo JF. Outcomes research and obstructive sleep apnea. Laryngoscope. 2000 Mar;110(3 Pt 3):16-20. doi: 10.1097/00005537-200003002-00005. PMID 10718409
- [Background] Temirbekov D, Gunes S, Yazici ZM, Sayin I. The Ignored Parameter in the Diagnosis of Obstructive Sleep Apnea Syndrome: The Oxygen Desaturation Index. Turk Arch Otorhinolaryngol. 2018 Mar;56(1):1-6. doi: 10.5152/tao.2018.3025. Epub 2018 Mar 1. PMID 29988275
- [Background] Rashid NH, Zaghi S, Scapuccin M, Camacho M, Certal V, Capasso R. The Value of Oxygen Desaturation Index for Diagnosing Obstructive Sleep Apnea: A Systematic Review. Laryngoscope. 2021 Feb;131(2):440-447. doi: 10.1002/lary.28663. Epub 2020 Apr 25. PMID 32333683
- [Background] Jacobowitz O, Schwartz AR, Lovett EG, Ranuzzi G, Malhotra A. Design and rationale for the treating Obstructive Sleep Apnea using Targeted Hypoglossal Nerve Stimulation (OSPREY) trial. Contemp Clin Trials. 2022 Aug;119:106804. doi: 10.1016/j.cct.2022.106804. Epub 2022 May 22. PMID 35613672
- [Background] Scharf MT. Reliability and Efficacy of the Epworth Sleepiness Scale: Is There Still a Place for It? Nat Sci Sleep. 2022 Dec 13;14:2151-2156. doi: 10.2147/NSS.S340950. eCollection 2022. PMID 36536636
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] De Meyer MMD, Vanderveken OM, De Weerdt S, Marks LAM, Carcamo BA, Chavez AM, Matamoros FA, Jacquet W. Use of mandibular advancement devices for the treatment of primary snoring with or without obstructive sleep apnea (OSA): A systematic review. Sleep Med Rev. 2021 Apr;56:101407. doi: 10.1016/j.smrv.2020.101407. Epub 2020 Nov 29. PMID 33326914
- [Background] Smith SS, Oei TP, Douglas JA, Brown I, Jorgensen G, Andrews J. Confirmatory factor analysis of the Epworth Sleepiness Scale (ESS) in patients with obstructive sleep apnoea. Sleep Med. 2008 Oct;9(7):739-44. doi: 10.1016/j.sleep.2007.08.004. Epub 2007 Oct 24. PMID 17921053
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Result] Hsu YB, Lan MY, Huang YC, Huang TT, Lan MC. The correlation between drug-induced sleep endoscopy findings and severity of obstructive sleep apnea. Auris Nasus Larynx. 2021 Jun;48(3):434-440. doi: 10.1016/j.anl.2020.09.018. Epub 2020 Oct 7. PMID 33039197